CLINICAL TRIAL: NCT06547957
Title: A First-in-Human Open-label, Phase I Dose Escalation and Expansion Cohort Study of EOS301984 as Monotherapy and in Combination With Other,Anticancer Treatments in Participants With Advanced Solid Tumors
Brief Title: A First-in-Human Study of EOS301984 as Monotherapy or Combination Therapy in Adult Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iTeos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APT-008; 2023-503844-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-28; First posted 2024-08-09 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors; neoplasm; cancer; phase I; immunotherapy; anticancer
MeSH Terms: conditions — Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1A dose escalation (Experimental): EOS301984 dose escalation as monotherapy
  Interventions: Drug: EOS301984
- Part 1B dose escalation (Experimental): EOS301984 in combination with other cancer therapies
  Interventions: Drug: EOS301984; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: EOS301984 — Multiple doses of EOS301984
  Other Names: EOS-984
Drug: Anti-PD-1 monoclonal antibody — Multiple doses of EOS301984 in combination with Anti-PD-1
  Arms: Part 1B dose escalation

SUMMARY:
APT-008 is an open-label, Phase I/Ib, dose escalation and expansion cohort study to evaluate the safety, tolerability, Pharmacokinetic (PK), Pharmacodynamic (PD), and preliminary efficacy of EOS301984 as monotherapy and in combination with other anticancer therapies in participants with advanced solid tumors.

ELIGIBILITY:
INCLUSION CRITERIA

* Provide a signed written informed consent before any study-specific evaluation.
* Be at least 18 years old on the day of signing informed consent.
* Have a histologically confirmed advanced solid tumor for which no standard approved treatment is available, or are ineligible for, or did not tolerate standard approved treatment.
* Have at least one tumor lesion measurable per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have adequate organ and marrow function.
* Agree to use adequate highly effective method of contraception during the study is mandatory, if Women of Childbearing Potential (WOCBP) or male.

EXCLUSION CRITERIA

* Have received prior systemic anticancer treatment including investigational agents within 4 weeks before the first dose of study treatment.
* Have major surgery planned or have had a major surgery within 5 weeks before the first dose of the study treatment.
* Have received prior radiotherapy within 2 weeks before the first dose of study treatment.
* Have allergy to study treatment(s) or any of its components.
* Have a history or current evidence of uncontrolled or significant cardiovascular disease. Unable to comply with the requirements of the study or who, in the opinion of the Investigator, should not participate in the study.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of EOS301984 alone and in combination with other anticancer agents in participants with advanced solid tumors | From first study treatment administration to last participant last follow-up (Up to 4 years)
Incidence and severity of AEs in patients receiving EEOS301984 | From first study treatment administration to last participant last follow-up (Up to 4 years)

SECONDARY OUTCOMES:
Mean and median Area under the curve (AUC) of EOS301984 following first dose and repeated administration at each dose level | From first dose up to 21 days repeated cycles
Mean and median Maximum concentration (Cmax) of EOS301984 following first dose and repeated administration at each dose level | From first dose up to 21 days repeated cycles
Define the recommended Phase 2 dose (RP2D) in participants with advanced tumors. | From first study treatment administration to last participant last follow-up (Up to 4 years)
Percentage of participants with Objective Response as determined by Investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | From first study treatment administration to last participant last follow-up (Up to 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Iteos Clinical Trials, Study Director — iTeos Therapeutics Inc.
Locations (6):
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - CHU de Liège, Liège
  - GZA Ziekenhuizen campus Sint-Augustinus, Wilrijk

IPD SHARING:
Plan to Share IPD: No